CLINICAL TRIAL: NCT03685149
Title: Pilot Randomized Trial With Flecainide in ARVC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Wojciech Zareba, Professor of Medicine/Cardiology, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00001910; R34HL143372 (NIH)
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: arrhythmogenic right ventricular cardiomyopathy; ARVC; Flecainide; ventricular arrhythmias; implantable cardioverter-defibrillator
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia | interventions — Flecainide

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blinded placebo-controlled crossover trial on the effect of flecainide on the frequency of ventricular arrhythmias of 38 ARVC patients. The crossover design requires a 10-week treatment with each patient receiving flecainide 100 mg bid and placebo for 4 weeks in a blinded randomized order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is double-blinded trial with all participants, investigators, and outcome assessors being blinded with except for the Data and Safety Monitoring Board (DSMB) members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flecainide (Active Comparator): The same subjects will be treated in a random order with flecainide or placebo for 4 weeks each with 1 week washout between crossover periods.
  Interventions: Drug: Flecainide Pill; Drug: Placebo
- Placebo (Placebo Comparator): The same subjects will be treated in a random order with flecainide or placebo for 4 weeks each with 1 week washout between crossover periods.
  Interventions: Drug: Flecainide Pill; Drug: Placebo

INTERVENTIONS:
Drug: Flecainide Pill — Flecainide pill or placebo 100 mg administered twice a day for 4 weeks each
  Other Names: Tambocor
Drug: Placebo — Flecainide pill or placebo 100 mg administered twice a day for 4 weeks each

SUMMARY:
Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is an inherited arrhythmia disorder with high risk of ventricular tachycardia or fibrillation, and implantable cardioverter defibrillator remains as therapy of choice. Antiarrhythmic therapy with different agents including beta-blockers, sotalol and amiodarone are usually not effective in reducing risk of arrhythmic events. Recent data indicated that flecainide effectively prevented the arrhythmias observed in the experimental ARVC animals and in small series of ARVC patients. These observations provide a strong rationale for conducting a pilot randomized clinical trial to determine whether flecainide will reduce ventricular arrhythmias in high-risk ARVC patients. This pilot study is designed as randomized double-blinded placebo-controlled crossover trial with administration of 100 mg of Flecainide or matching placebo twice a day for 4 weeks each with a washout period.

Primary specific aim of this pilot trial is to determine whether Flecainide administration is associated with a significant reduction of number of ventricular ectopic beats (VEBs) in ARVC patients with implantable cardioverter-defibrillator (ICD).

DETAILED DESCRIPTION:
Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC) is an inherited arrhythmia disorder with high risk of ventricular tachycardia or fibrillation, and implantable cardioverter defibrillator remains as therapy of choice. Antiarrhythmic therapy with different agents including beta-blockers, sotalol and amiodarone are usually not effective in reducing risk of arrhythmic events. Recent data indicated that flecainide effectively prevented the arrhythmias observed in the experimental ARVC animals and in small series of ARVC patients. These observations provide a strong rationale for conducting a pilot randomized clinical trial to determine whether flecainide will reduce ventricular arrhythmias in high-risk ARVC patients. This pilot study is designed as randomized double-blinded placebo-controlled crossover trial with administration of 100 mg of Flecainide or matching placebo twice a day for 4 weeks each with a washout period.

Primary specific aim of this pilot trial is to determine whether Flecainide administration is associated with a significant reduction of number of ventricular ectopic beats (VEBs) in ARVC patients with implantable cardioverter-defibrillator (ICD).

Secondary specific aims are:

1. to assess safety of flecainide administration with particular emphasis on proarrhythmic response measured by:

   1. VEBs on ECG monitoring,
   2. nonsustained and sustained ventricular tachycardia (VT) or ventricular fibrillation (VF) episodes documented on ICD interrogation, and
   3. effects of Flecainide on QRS morphology and duration.
2. to assess effects of flecainide on burden of VT runs in 7-day ECG recordings.
3. to assess effects of flecainide on burden of atrial premature beats in 7-day recordings.
4. to demonstrate feasibility of enrollment of rare inherited arrhythmia ARVC patients in a randomized study in the light of planned future large clinical trial with VT/VF/death as endpoint.

Study population will include 38 ARVC patients diagnosed with the 2010 ARVC Task Force Criteria who are at least 18 years old, have implanted ICD, and show at least 500 VEBs in a 24-hour Holter recording. Patients on other pharmacological antiarrhythmic treatment other than beta-blockers and patients with prior catheter VT ablation will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Subjects who have been diagnosed with ARVC and meet 2010 Modified Task Force Criteria for ARVC as affected.
* At minimum 500 VEBs on the most recent 24-hour Holter monitor recording prior to consent or after consent if a subsequent recording is required after 5 day washout following discontinuation of anti-arrhythmic medication.
* Functioning implanted cardioverter defibrillator with remote interrogation capability.
* Subjects should be on a beta-blocker including metoprolol, propranolol, atenolol, nadolol, carvedilol or bisoprolol unless contraindication to beta-blockers exists.
* Persons prescribed quinidine, procainamide, propafenone, disopyramide, dronedarone phenytoin, mexiletene, flecainide, may be included after 5 day washout period with subsequent 24 Hour Holter obtained after washout period.
* Persons prescribed sotalol must be included after 5 day washout period during which another beta-blocker may be administered with subsequent 24 Hour Holter obtained.
* Subject and personal physician and or cardiologist must agree not to use any antiarrhythmic medications during the 10 weeks of participation, unless needed for management of life-threatening arrhythmias.
* All subjects must agree to use medically acceptable contraceptive measures during participation unless documented as surgically sterile or post-menopausal (no menstrual periods for more than one year).

Exclusion Criteria:

* Prescribed amiodarone or dofetilide at the time of consent.
* Left ventricular ejection fraction ≤40% by any imaging modality: echocardiography, angiography, cardiac magnetic resonance imaging (CMRI), or cardiac nuclear test on the most recent test.
* New York Heart Association (NYHA) heart failure class III or IV at time of consent.
* Prior myocardial infarction at any time in the past.
* Pacemaker dependent rhythm at the time of consent.
* Renal impairment (GFR <30 mL/min/m2).
* Prior diagnosis of severe hepatic impairment.
* Pregnant or plan to become pregnant during the course of the trial (Flecainide has not been adequately studied in pregnant women). Pregnancy test is required for women of child-bearing potential prior to randomization.
* Participating in any other interventional clinical trial.
* Unwilling or unable to cooperate with the protocol.
* Lives at such a distance from the clinic that travel for the consent visit would be unusually difficult.
* Decisionally impaired adults, those of questionable capacity, those who cannot manage taking the study drug per the prescribed regimen, and those who cannot consent for themselves will not be recruited for this study.
* Unwilling to sign the consent for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Zareba, MD, PhD, Principal Investigator — University of Rochester
Locations (6):
- United States (6):
  - University of Colorado, Denver, Colorado
  - John Hopkins University, Baltimore, Maryland
  - New York University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - University of Pensylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
This is a small pilot trial with limited dataset which will be mostly explored by enrolling center investigators.

REFERENCES:
- [Background] Marcus FI, Zareba W, Calkins H, Towbin JA, Basso C, Bluemke DA, Estes NA 3rd, Picard MH, Sanborn D, Thiene G, Wichter T, Cannom D, Wilber DJ, Scheinman M, Duff H, Daubert J, Talajic M, Krahn A, Sweeney M, Garan H, Sakaguchi S, Lerman BB, Kerr C, Kron J, Steinberg JS, Sherrill D, Gear K, Brown M, Severski P, Polonsky S, McNitt S. Arrhythmogenic right ventricular cardiomyopathy/dysplasia clinical presentation and diagnostic evaluation: results from the North American Multidisciplinary Study. Heart Rhythm. 2009 Jul;6(7):984-92. doi: 10.1016/j.hrthm.2009.03.013. Epub 2009 Mar 11. PMID 19560088
- [Background] Marcus FI, McKenna WJ, Sherrill D, Basso C, Bauce B, Bluemke DA, Calkins H, Corrado D, Cox MG, Daubert JP, Fontaine G, Gear K, Hauer R, Nava A, Picard MH, Protonotarios N, Saffitz JE, Sanborn DM, Steinberg JS, Tandri H, Thiene G, Towbin JA, Tsatsopoulou A, Wichter T, Zareba W. Diagnosis of arrhythmogenic right ventricular cardiomyopathy/dysplasia: proposed modification of the task force criteria. Circulation. 2010 Apr 6;121(13):1533-41. doi: 10.1161/CIRCULATIONAHA.108.840827. Epub 2010 Feb 19. PMID 20172911
- [Background] Corrado D, Link MS, Calkins H. Arrhythmogenic Right Ventricular Cardiomyopathy. N Engl J Med. 2017 Jan 5;376(1):61-72. doi: 10.1056/NEJMra1509267. No abstract available. PMID 28052233
- [Background] Cerrone M, Montnach J, Lin X, Zhao YT, Zhang M, Agullo-Pascual E, Leo-Macias A, Alvarado FJ, Dolgalev I, Karathanos TV, Malkani K, Van Opbergen CJM, van Bavel JJA, Yang HQ, Vasquez C, Tester D, Fowler S, Liang F, Rothenberg E, Heguy A, Morley GE, Coetzee WA, Trayanova NA, Ackerman MJ, van Veen TAB, Valdivia HH, Delmar M. Plakophilin-2 is required for transcription of genes that control calcium cycling and cardiac rhythm. Nat Commun. 2017 Jul 24;8(1):106. doi: 10.1038/s41467-017-00127-0. PMID 28740174
- [Background] Ermakov S, Gerstenfeld EP, Svetlichnaya Y, Scheinman MM. Use of flecainide in combination antiarrhythmic therapy in patients with arrhythmogenic right ventricular cardiomyopathy. Heart Rhythm. 2017 Apr;14(4):564-569. doi: 10.1016/j.hrthm.2016.12.010. Epub 2016 Dec 9. PMID 27939893

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 7 enrolling sites in the study. Recruitment took place at 6 enrolling sites between July 23, 2019 and May 2, 2022.
Groups:
- Placebo, Then Flecainide: Participants first received Placebo pill (matching Flecainide 100 mg) twice a day for 4 weeks. After a washout period of 1 week, they then received Flecainide pill (100 mg) twice a day for 4 weeks with subsequent 1 week of washout.
- Flecainide, Then Placebo: Participants first received Flecainide pill (100 mg) twice a day for 4 weeks. After a washout period of 1 week, they then received Placebo pill (matching Flecainide 100 mg) twice a day for 4 weeks, with subsequent 1 week of washout.
Period: First Intervention (4 Weeks)
Arm/Group | Placebo, Then Flecainide | Flecainide, Then Placebo
Started | 11 | 11
Completed | 10 | 9
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (1 Week)
Arm/Group | Placebo, Then Flecainide | Flecainide, Then Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Placebo, Then Flecainide | Flecainide, Then Placebo
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Flecainide | Flecainide, Then Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 43 (14) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Ventricular Ectopic Beats (VEBs) Per Day
Description: Number of ventricular ectopic beats (VEBs) per day in a 7-day ECG recording
Time Frame: 7-day period
Population: 18 subjects had ECG recordings on placebo and 18 had on flecainide, with 2 recordings missing, 17 subjects had both recordings
Measure: Median (Inter-Quartile Range); unit: number of VEBs per day
Groups:
- Placebo; Flecainide: Per randomization: 1) Participants first received Placebo pill (matching Flecainide 100 mg) twice a day for 4 weeks. After a washout period of 1 week, they then received Flecainide pill (100 mg) twice a day for 4 weeks with subsequent 1 week of washout.
  or 2) Participants first received Flecainide pill (100 mg) twice a day for 4 weeks. After a washout period of 1 week, they then received Placebo pill (matching Flecainide 100 mg) twice a day for 4 weeks, with subsequent 1 week of washout.
Arm/Group | Placebo | Flecainide
Number analyzed (Participants) | 18 | 18
number of VEBs per day | 2685 [1187 to 5431] | 677 [310 to 1663]
Statistical Analysis 1: Comparison: Placebo vs Flecainide; Test type: Superiority; p < 0.0001, Mixed Models Analysis; percent reduction = 72, 95% CI 2-sided [56 to 82]

2. Secondary Outcome: Number of Participants With Proarrhythmic Response to Flecainide
Description: Nonsustained and sustained ventricular tachycardia and ventricular fibrillation recorded by implantable cardioverter-defibrillator (ICD) during 4-week treatment periods.
Time Frame: 4 weeks
Population: 19 subjects had data regarding ICD-documented arrhythmias
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Flecainide
Number analyzed (Participants) | 19 | 19
Participants | 3 | 3
Statistical Analysis 1: Comparison: Placebo vs Flecainide; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0

3. Secondary Outcome: Ventricular Tachycardia (VT) Burden
Description: Number of VT runs/episodes recorded per day on a 7-day ECG recording
Time Frame: 7-day period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of VTs per day
Arm/Group | Placebo | Flecainide
Number analyzed (Participants) | 18 | 18
number of VTs per day | 0.4 (0.5) | 0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Flecainide; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Atrial Premature Beats (APBs) Per Day
Description: Number of atrial premature beats (APBs) per day in a 7-day ECG recording
Time Frame: 7-day period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of APBs per day
Arm/Group | Placebo | Flecainide
Number analyzed (Participants) | 18 | 18
number of APBs per day | 32 [4 to 102] | 8 [1 to 61]
Statistical Analysis 1: Comparison: Placebo vs Flecainide; Test type: Superiority; p = 0.207, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 weeks on Flecainide and 4 weeks on matching Placebo in this cross-over study
Arm/Group | Placebo | Flecainide
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/22
Other Adverse Events (participants affected / at risk) | 7/22 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Flecainide (N=22)
Ventricular tachycardia requiring implantabale cardioverter defibrillator (ICD) therapy (Cardiac disorders) | 1 (2) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Flecainide (N=22)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03685149/Prot_SAP_000.pdf